CLINICAL TRIAL: NCT04912713
Title: Influencia Del Estrés Agudo en el Aprendizaje Motor de Una Tarea Manual Precisa y en la Capacidad de Imaginación Motora
Brief Title: Influence of Acute Stress on Motor Learning and Motor Imagery Ability in Young Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susana Nunez Nagy (Other)
Collaborators: University of Alcala (Other); Universidad Complutense de Madrid (Other); European University of Madrid (Other); Claude Bernard University (Other)
Responsible Party: Sponsor-Investigator, Susana Nunez Nagy, PhD. Associate Professor of Physiotherapy, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CEID2022/2/036
Record Dates: First submitted 2021-05-26; First posted 2021-06-03 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Stress, Psychological
Keywords: Stress, Psychological; Learning; Memory; Movement
MeSH Terms: conditions — Stress, Psychological | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: As participants complete the State-Trait Anxiety Inventory, and are found to be free of trait anxiety, and state anxiety, they will be randomised in parallel to one of the two intervention groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant does not know what the other participants are doing, the researcher knows which study and group the subject is in, but only sets up the computerized presentations for each group and assigns folders within the computer that collects the data, thus avoiding a possible information bias, and finally, another researcher blind to the intervention will analyse the data to obtain the results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): This group will be randomly immersed in ice water (2°C temperature) for preset times and instructed to remove their hand if they cannot withstand these times. In total there will be 5 attempts with durations of 90, 60, 60, 60, 90 and 60 s respectively. Between dive attempts they will be instructed to put their arm on a towel and immediately do the arithmetic task of counting backwards from the number 2043 as quickly and accurately as they can. Each time they make a mistake in the mental task, they will be given negative feedback and must start again from the number 2043. The duration of the 4 arithmetic tasks (between each of the 5 immersion attempts) will be fixed at 45, 60, 90 and 45 s respectively.
  Interventions: Other: Stress group
- Arm 2 (Active Comparator): This group will not be falsely recorded or evaluated. They will be randomly immersed in warm water (35-37°C temperature) for preset times and instructed to remove their hand if they cannot withstand these times. In total there will be 5 attempts with durations of 90, 60, 60, 60, 90 and 60 s respectively. Between dive attempts they will be instructed to put their arm on a towel and immediately do the simple counting task, in which they will have to count consecutively from 1 to 25 at their own pace. If they reach 25 they must start again and will never be given negative feedback. The duration of the 4 arithmetic tasks (between each of the 5 immersion attempts) will be fixed at 45, 60, 90 and 45 s respectively
  Interventions: Other: Control group

INTERVENTIONS:
Other: Stress group — This group will perform the MAST stress protocol
  Arms: Arm 1
Other: Control group — This group will perform the MAST control protocol
  Arms: Arm 2

SUMMARY:
In motor learning, it is essential to consider that movements are produced by the cooperation and combination of many brain structures and are influenced by the emotions to which individuals are subjected. Several neural circuits have been identified that closely link the emotional system and the motion control system.

Stress is a physiological or psychological response to internal or external stressors. In principle, it has an adaptive role. However, the neuroendocrine and autonomic response generated by stress can affect cognitive processes such as memory. In addition, it has been shown to influence motor learning, especially the execution of skills in the early stages of learning.

Understanding how movement, emotions and interactions are regulated is significant because of the large number of movements humans perform. Of these, manual tasks represent precise movements that require the integration of many elements by the nervous system to perform these tasks successfully. It is still unknown how acute stress influence the way manual tasks are learned.

On the other hand, motor imagery (MI) is a cognitive process that is an important contributor to how movements are planned and executed. Its use has been recommended to improve movement learning and task execution. For an MI program to be effective and individualized, it is imperative to know this ability. However, it is also still unknown how acute stress can affect our motor imagery ability.

The main objective of this study is to determine and quantify the effects of acute stress in the learning of a precise manual task not previously trained on four parameters of fine motor control: trajectory error, timing error, timing accuracy, and task accuracy. On the other hand, the aim is to determine if the capacity of internal visual, external visual, and kinesthetic imagery, and the temporal congruence between movement execution and imagery varies when we are subjected to acute stress.

It is expected that non-anxious, non-stressed participants who are not induced with acute stress will show better motor performance on the fine motor task and better motor imagery ability and temporal congruence. In contrast, it is expected that participants without anxiety and stress who are induced with acute stress will show poorer motor performance on the fine motor task, and poorer motor imagery ability and temporal congruence.

DETAILED DESCRIPTION:
In order to meet the study objectives of determining and quantifying the effects of acute stress on learning a precise manual task and on motor imagery ability, this study will be conducted. The development of the study will take place in a conditioned room belonging to the University of Alcalá, the Complutense University of Madrid, the European University of Madrid, or Claude Bernard University Lyon 1. The study may also be carried out in other Spanish and international university centers, subject to the consent and permission of the respective centres. The study will be carried out by all national and international laws, regulations, and recommendations.

The study design will be longitudinal, experimental, randomized, and double-blind, as specified in the present registry.

The study population will be composed of participants who are undergraduate and postgraduate students at the university centers where the study will be carried out, from which they will be recruited. All participants included in the study must meet the study selection criteria and participate voluntarily after reading the information sheet and signing the informed consent form.

The study will consist of two intervention groups, in which the Maastricht Acute Stress Test (MAST) protocol will be performed: one group will perform the acute stress induction protocol (MAST stress) and the other group will perform the no stress induction control protocol (MAST control). Each group will consist of a minimum number of 30 subjects to be able to study the desired effect.

After each participant freely chooses to participate in the study, an initial questionnaire will be administered to ensure that they meet the criteria for inclusion in the study. At this point, they will be coded by assigning them a number, which will serve to identify each participant throughout the study. Participants will take the State-Trait Anxiety Inventory (STAI), one of the most widely used instruments for the self-reported assessment of anxiety and equivalent to a measure of stress, as it considers the amount of stressful stimulus. Thus, the two components of anxiety will be assessed: state anxiety and trait anxiety. Participants with scores indicative of state or trait anxiety will be excluded from the study, and those with scores indicating neither trait anxiety nor state anxiety will be included. Included participants will be randomized through sealed envelopes stratified by gender to one of two experimental groups: MAST stress, or MAST control. They will also take the Edinburgh Handedness Inventory (EHI) to determine the participant's laterality, and the Movement Imagery Questionnaire-3 (MIQ-3) to measure internal visual, external visual, kinaesthetic imagery capacity. At the same time of MIQ-3, the experimenter will record the execution and imagery times were recorded (for subsequent calculation of the time discrepancy between executed and imagery as a measure of temporal congruence between them). Depending on the group to which they have been assigned, they will perform the corresponding MAST protocol (stress or control). MAST stress is a non-invasive protocol to induce acute stress in the laboratory that combines components of psychological stress (evaluative social threat, uncontrollability, and unpredictability) and physical stress (sensation of pain through intense cold). The MAST control is a homologous protocol to the stress protocol but has no psychological or physical stressor components. After MAST protocol, participants will learn a precise manual task with the non-dominant hand. The task will consist of going over a 127 mm circumference on a graphics tablet at a rate of 2 seconds per lap, which will be set by a metronome using a wireless pen that will leave no trace of ink but will store the data in the MATLAB program via the graphics tablet. Thus, data from the acquisition and short-term retrieval of the task will be recorded. Afterward, there will be a 20-minute break during which participants will perform the MIQ-3 and the experimenter will record the execution and imagery times again. Finally, the task data will be collected to record the long-term retrieval of the manual task.

In addition, during all experiments, electrodermal activity and heart rate variability will be recorded using the Empatica E4 physiological variable measurement wristband. This measurement of physiological variables will serve to confirm that a significant emotional effect has been generated and to test motor imagery processes since both acute stress and motor imagery produce activation of the autonomic nervous system.

The analysis and processing of data from MATLAB version R2020b, and the Empatica E4 wristband will be performed using RStudio software and Kubios HRV software (for HRV analysis).

First, appropriate statistical analyses will be performed to see if the data are distributed according to a standard curve through the Shapiro-Wilk test and to assess the influence of sex and age.

Subsequently, the descriptive analysis of the relative and absolute frequencies for the qualitative variables of gender and age will be carried out, and their homogeneity will be tested using the Chi-square test. The descriptive analysis of the quantitative variables of trajectory error, timing error, timing accuracy, task accuracy, electrodermal activity, heart rate variability, kinaesthetic, internal visual, and external visual imagery, and discrpenacy times will also be carried out. If the variable conforms to the normal, the mean, range, and standard deviation shall be calculated. If it does not conform to the normal, non-parametric tests will be performed.

Comparative analysis will be performed using mixed ANOVA to see the differences in the mean values respective to motor control (trajectory error, timing error, timing accuracy, and task accuracy). A further ANOVA analysis will take place for imagery ability and discrepancy times, comparing the results obtained at the two respective points during the experiment.

The effect of learning between laps will be analyzed by repeated-measures ANOVA comparing each motor control measurement parameter with respect to the lapping factor. Electrodermal activity, and heart rate variability during the measurement of imagery ability, emotional state induction, manual task acquisition, and its retrieval in the short and long term will also be studied by repeated-measures ANOVA.

For hypothesis testing, a significance level of 0.05 will be set.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 35 years of age.
* Normal or corrected vision specifying the method of correction.
* Normal or corrected hearing specifying method of correction.
* Unfamiliar with the assessment and uses of motor imagery.

Exclusion Criteria:

* Subjects who have suffered fractures, dislocations, or traumatic processes in any segment of the non-dominant upper limb or fingers, wrist, or elbow of the dominant upper limb in the last 6 months.
* Subjects with learning disabilities or problems in reading or writing.
* Subjects with a history of any neurological disease, cardiovascular disease, myopathic disease, epileptic seizure, absence seizure, sleep apnoea, chronic fatigue syndrome, or fibromyalgia.
* Taking any medication to suppress anxiety, to sleep, antidepressants, antihistamines, muscle relaxants, psychotropic, or other medications that interfere with the nervous system.
* Intake of nervous system depressants or stimulants such as caffeine or theine in the last 8 hours.
* Presence of State-Trait Anxiety Inventory scores corresponding to trait anxiety and state anxiety.
* Presence of localised skin lesion or disease in the wrist area.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Trayectory error | During manual task performance in acquisition, short-term retrieval, and long-term retrieval.
  It shall be the sum of the error between each of the points defining the path of the circumference. Pixels squared shall be considered as the unit of length measurement. To be recorded and measured with MATLAB. To be recorded and measured with MATLAB.
Timing error | During manual task performance in acquisition, short-term retrieval, and long-term retrieval.
  It is the absolute value of the difference between the duration of 2 seconds requested from the subjects and the total time elapsed in the execution of the trajectory. It shall be expressed in seconds (s). It shall be recorded and measured using MATLAB.
Timing accuracy | During manual task performance in acquisition, short-term retrieval, and long-term retrieval.
  The ability of the subject to learn the task at the requested rate of 2 seconds per lap. It shall be expressed in square pixels per second. It shall be recorded and measured by MATLAB.
Task accuracy | During manual task performance in acquisition, short-term retrieval, and long-term retrieval.
  It shall be the ability of the subject to learn at any rate. It shall be expressed in pixels per second. It shall be recorded and measured by MATLAB.
Motor Imagery Capacity | Before induction of acute stress and in the resting period between short-term and long-term retrieval after induction of acute stress.
  This will be measured using the Movement Imagery Questionnaire-3, differentiating between the kinaesthetic, external visual and internal visual imagination subscales, each scored on a Likert scale from 1 to 7.
Discrepancy time | Before induction of acute stress and in the resting period between short-term and long-term retrieval after induction of acute stress.
  It will be the difference between the execution times and imagery of the MIQ-3 items. It will be measured with a stopwatch by the experimenter.

SECONDARY OUTCOMES:
Electrodermal Activity. | During the procedure
  The skin conductance level shall be analyzed in terms of tonic Electrodermal Activity. It shall be recorded and measured by Empatica E4 wristband.
Heart Rate Variability. | During the procedure
  It will be analysed in the frequency domain, in its low and high frequency bands and in the ratio between them. It shall be recorded and measured by Empatica E4 wristband.

CONTACTS AND LOCATIONS:
Overall Officials: Sara T Trapero Asenjo, Master, Principal Investigator — University of Alcala; Susana N Núñez Nagy, PhD, Study Director — University of Alcala; Sara F Fernández Guinea, PhD, Study Director — Universidad Complutense de Madrid
Locations (4):
- Claude Bernard University Lyon 1, Villeurbanne, Auvergne-Rhône-Alpes, France
- Spain (3):
  - University of Alcala, Alcalá de Henares, Madrid
  - Complutense University of Madrid, Pozuelo de Alarcón, Madrid
  - European University of Madrid, Villaviciosa de Odón, Madrid

REFERENCES:
- [Background] Coombes SA, Cauraugh JH, Janelle CM. Emotion and movement: activation of defensive circuitry alters the magnitude of a sustained muscle contraction. Neurosci Lett. 2006 Apr 3;396(3):192-6. doi: 10.1016/j.neulet.2005.11.048. Epub 2005 Dec 20. PMID 16376016
- [Background] Ahn SN, Lee J. Effects of sensory awareness, imagery and observation on electroencephalography in adult with psychological stress. J Phys Ther Sci. 2019 Jan;31(1):17-19. doi: 10.1589/jpts.31.17. Epub 2019 Jan 10. PMID 30774198
- [Background] MacIntyre TE, Madan CR, Moran AP, Collet C, Guillot A. Motor imagery, performance and motor rehabilitation. Prog Brain Res. 2018;240:141-159. doi: 10.1016/bs.pbr.2018.09.010. Epub 2018 Oct 24. PMID 30390828
- [Background] Schuster C, Hilfiker R, Amft O, Scheidhauer A, Andrews B, Butler J, Kischka U, Ettlin T. Best practice for motor imagery: a systematic literature review on motor imagery training elements in five different disciplines. BMC Med. 2011 Jun 17;9:75. doi: 10.1186/1741-7015-9-75. PMID 21682867
- [Background] Trapero-Asenjo S, Gallego-Izquierdo T, Pecos-Martin D, Nunez-Nagy S. Translation, cultural adaptation, and validation of the Spanish version of the Movement Imagery Questionnaire-3 (MIQ-3). Musculoskelet Sci Pract. 2021 Feb;51:102313. doi: 10.1016/j.msksp.2020.102313. Epub 2020 Dec 9. PMID 33310512
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Smeets T, Cornelisse S, Quaedflieg CW, Meyer T, Jelicic M, Merckelbach H. Introducing the Maastricht Acute Stress Test (MAST): a quick and non-invasive approach to elicit robust autonomic and glucocorticoid stress responses. Psychoneuroendocrinology. 2012 Dec;37(12):1998-2008. doi: 10.1016/j.psyneuen.2012.04.012. Epub 2012 May 18. PMID 22608857
- [Background] Bali A, Jaggi AS. Clinical experimental stress studies: methods and assessment. Rev Neurosci. 2015;26(5):555-79. doi: 10.1515/revneuro-2015-0004. PMID 26020552